CLINICAL TRIAL: NCT02077335
Title: Phase II Study of High-dose Rate (HDR) Monotherapy for the Treatment of Low and Intermediate Risk Prostate Cancer
Brief Title: Study of High-dose Rate (HDR) Monotherapy for Low and Intermediate Risk Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSSS de Gatineau (Other)
Responsible Party: Principal Investigator, Marc Gaudet, Radiation Oncologist, CSSS de Gatineau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSSSG-001
Record Dates: First submitted 2014-02-23; First posted 2014-03-04 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: Brachytherapy; Monotherapy; HDR
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HDR brachytherapy monotherapy (Experimental): Radiation therapy: Treatment with 2 separate HDR brachytherapy implants, each with one fraction of 13.5 Gray (Gy) with an interval of 7-14 days between treatments.
  Interventions: Radiation: HDR brachytherapy monotherapy

INTERVENTIONS:
Radiation: HDR brachytherapy monotherapy — Radiation therapy in the study consists of treatment with 2 separate interstitial HDR brachytherapy procedures with temporary interstitial catheters, each with one fraction of 13.5 Gray (Gy). Both procedures will be done in an identical manner. The 2 procedures will be separated by an interval of 7-14 days Treatments will be done with interstitial catheters inserted transperineally with transrectal ultrasound guidance under sterile conditions. Optimization of treatment plan will be done with Brachyvision software (Varian, Palo Alto CA) based on CT-scan imaging done post-implant. Optimization parameters will be the following:
  Prostate :
  * V100 > 95%
  * V150 30-35%
  * V200 < 15%
  * D90 > 90% (12,15Gy)
  Bladder
  • V75 < 1cc
  Rectum
  • V75 < 1cc
  Urethra
  V125 = 0cc D10 < 120%
  Treatments will be carried out with an Iridium-192 afterloader. Source and all catheters will be removed from the patient at the end of the procedure.

SUMMARY:
The purpose of this study is to determine the clinical efficacy and toxicity of High-dose rate (HDR) brachytherapy as monotherapy for the treatment of low risk and intermediate risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven Adenocarcinoma of the Prostate
* Clinical stage T1c, T2a or T2b
* PSA less than 20 ng/ml
* Gleason Score 6 or 7

Exclusion Criteria:

* Age less than 18 years
* Clinical stage T2c, T3 ou T4
* Clinical Stage N1
* Clinical Stage M1
* Prostate Specific Antigen (PSA) more than 20 ng/ml
* Gleason score 8 or higher
* IPSS score 19 or higher with alpha-blockers
* Past radiation therapy to the pelvis
* History of Collagen Vascular Disease
* History of Inflammatory Bowel Disease
* Bilateral Hip Prosthesis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
  Disease free survival as evaluated by absence of biochemical recurrence (Phoenix criteria) and absence of clinically/radiologically diagnosed local, regional or distant recurrence.

SECONDARY OUTCOMES:
Genito-urinary (GU) toxicity | 6 weeks, 2 years and 5 years post treatment
  Toxicity according to International prostate symptom score (IPSS) and Expanded Prostate Index Composite (EPIC) questionnaires.

OTHER OUTCOMES:
Overall survival | 5 years
Gastro-Intestinal (GI) Toxicity | 6 weeks, 2 years and 5 years post treatment
  Toxicity according to Expanded Prostate Index Composite (EPIC) questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- CSSS de Gatineau, Gatineau, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No